CLINICAL TRIAL: NCT07090161
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Iloperidone for the Treatment of Participants With Uncontrolled Hypertension
Brief Title: Evaluation of Efficacy and Safety of Iloperidone for the Treatment of Participants With Uncontrolled Hypertension
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VP-VYV-683-2401
Record Dates: First submitted 2025-07-22; First posted 2025-07-29 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Hypertension; Uncontrolled Hypertension
Keywords: iloperidone; hypertension; uncontrolled hypertension
MeSH Terms: conditions — Hypertension | interventions — iloperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental/Iloperidone (Experimental)
  Interventions: Drug: iloperidone
- Placebo Comparator (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: iloperidone — iloperidone
  Other Names: Fanapt
  Arms: Experimental/Iloperidone
Drug: Placebo — placebo comparator
  Arms: Placebo Comparator

SUMMARY:
A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Iloperidone for the Treatment of Participants with Uncontrolled Hypertension

ELIGIBILITY:
Inclusion Criteria:

* SiSBP >/= 130 mmHg despite >8 weeks treatment w/ 1 or more antihypertensive therapies

Exclusion Criteria:

* Confirmed Grade 3/severe hypertension (SiSBP >/= 180 mmHg, SiDBP >/= 120 mmHg), unstable cardiac disease, renal insufficiency

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to treatment week 4 in SiSBP | screening to treatment week 4

CONTACTS AND LOCATIONS:
Locations (28):
- United States (28):
  - Vanda Investigative Site, Phoenix, Arizona
  - Vanda Investigative Site, Tempe, Arizona
  - Vanda Investigative Site, Tucson, Arizona
  - Vanda Investigative Site, Chula Vista, California
  - Vanda Investigative Site, Dublin, California
  - Vanda Investigative Site, Valencia, California
  - Vanda Investigative Site, Walnut Creek, California
  - Vanda Investigative Site, Doral, Florida
  - Vanda Investigative Site, Fort Myers, Florida
  - Vanda Investigative Site, Columbus, Georgia
  - Vanda Investigative Site, Oak Brook, Illinois
  - Vanda Investigative Site, Tinley Park, Illinois
  - Vanda Investigative Site, El Dorado, Kansas
  - Vanda Investigative Site, Wichita, Kansas
  - Vanda Investigative Site, Lexington, Kentucky
  - Vanda Investigative Site, Hazelwood, Missouri
  - Vanda Investigative Site, Las Vegas, Nevada
  - Vanda Investigative Site, Mount Kisco, New York
  - Vanda Investigative Site, Rochester, New York
  - Vanda Investigative Site, Kinston, North Carolina
  - Vanda Investigative Site, Cincinnati, Ohio
  - Vanda Investigative Site, Norman, Oklahoma
  - Vanda Investigative Site, Oklahoma City, Oklahoma
  - Vanda Investigative Site, Charleston, South Carolina
  - Vanda Investigative Site, Carrollton, Texas
  - Vanda Investigative Site, Salt Lake City, Utah
  - Vanda Investigative Site, Burke, Virginia
  - Vanda Investigative Site, Norfolk, Virginia